CLINICAL TRIAL: NCT00504660
Title: Combination of 6-Thioguanine, Capecitabine, Celecoxib and Temozolomide or CCNU for Recurrent Anaplastic Glioma and Glioblastoma Multiforme
Brief Title: 6-TG, Capecitabine and Celecoxib Plus TMZ or CCNU for Anaplastic Glioma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0600
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Anaplastic Glioma of Brain; Glioblastoma Multiforme; Brain Cancer
Keywords: Anaplastic Glioma; Glioblastoma Multiforme; Brain Cancer; 6-Thioguanine; Capecitabine; Celecoxib; Temozolomide; Xeloda; Temodar; TMZ; CCNU; 6-TG
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Capecitabine; Celecoxib; Temozolomide; Lomustine; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: Anaplastic Tumors (Active Comparator): Anaplastic Tumors - 6-TG 80 mg/m^2 orally (PO) every 6 hours Day 1-3; Temozolomide 150 mg/m^2 PO daily Days 4-8, after 6 day rest Capecitabine 825 mg/m^2 and Celebrex 400 mg PO every 12 hours Day 14-27 for 28 day course.
  Interventions: Drug: Capecitabine; Drug: Celecoxib (Celebrex); Drug: Temozolomide; Drug: 6-Thioguanine
- 2: Anaplastic Tumors (Active Comparator): Anaplastic Tumors - 6-TG 80 mg/m^2 PO every 6 hours Day 1-3, Lomustine 100 mg/m^2 PO on Day 4; Capecitabine 825 mg/m^2 PO every 12 hours Days 11-24, and Celebrex 400 mg PO every 12 hours Days 11-24.
  Participants if previously received Temozolomide but not Lomustine (CCNU) will receive Lomustine; or if had Gliadel wafers and Temozolomide with radiotherapy (XRT) will receive Temozolomide.
  Interventions: Drug: Capecitabine; Drug: Celecoxib (Celebrex); Drug: Lomustine; Drug: 6-Thioguanine
- 3: Glioblastoma Multiforme (Active Comparator): Glioblastoma Multiforme - 6-TG 80 mg/m^2 PO every 6 Hours Day 1-3; Capecitabine 825 mg/m^2 PO every 12 hours Days 14-27 and Celebrex 400 mg PO every 12 hours Day 11-24; Temozolomide 150 mg/m^2 PO daily Days 4-8 OR CCNU (Lomustine) 100 mg/m2 orally Day 4 of each 42-day cycle.
  Participants receive Temozolomide if not had previous treatment and if had prior CCNU. Those previously treated with Temozolomide but not CCNU receive CCNU, and those that had Gliadel and Temozolomide with XRT receive Temozolomide.
  Interventions: Drug: Capecitabine; Drug: Celecoxib (Celebrex); Drug: Temozolomide; Drug: Lomustine; Drug: 6-Thioguanine

INTERVENTIONS:
Drug: Capecitabine — Arms 1,3 = 825 mg/m^2 By Mouth (PO) Every 12 Hours on Day 14-27; Arms 2,3 = 825 mg/m^2 PO Every 12 Hours on Day 11-24.
  Other Names: Xeloda
Drug: Celecoxib (Celebrex) — Arms 1,3 = 400 mg PO Every 12 Hours On Day 14-27; Arms 2,3 = 400 mg PO Every 12 Hours On Day 11-24.
  Other Names: Celebrex
Drug: Temozolomide — Arms 1,3 = 150 mg/m^2 PO Daily On Day 4-8.
  Other Names: Temodar; TMZ
  Arms: 1: Anaplastic Tumors; 3: Glioblastoma Multiforme
Drug: Lomustine — Arms 2,3 = 100 mg/m^2 PO on Day 4.
  Other Names: CCNU
  Arms: 2: Anaplastic Tumors; 3: Glioblastoma Multiforme
Drug: 6-Thioguanine — Arms 1,2,3 = 80 mg/m^2 PO Every 6 Hours on Day 1-3.
  Other Names: Thioguanine; 6-TG

SUMMARY:
The goal of this clinical research study is to learn if the combination of 6-Thioguanine, Xeloda (capecitabine), and Celebrex (celecoxib) with Temodar (temozolomide) or Lomustine (CCNU) is effective in the treatment of recurrent or progressive anaplastic glioma or glioblastoma multiforme in patients who have failed previous treatments. The safety of these combination treatment will also be studied.

Objectives:

1.1 To determine the efficacy, as measured by 12 month progression-free survival, of TEMOZOLOMIDE or CCNU with 6-THIOGUANINE followed by CAPECITABINE and CELECOXIB in the treatment of patients with recurrent and/or progressive anaplastic gliomas or glioblastoma multiforme.

1.2 To determine the long-term toxicity of TEMOZOLOMIDE or CCNU with 6-THIOGUANINE followed by CAPECITABINE and CELECOXIB in recurrent anaplastic glioma or glioblastoma multiforme patients treated in this manner.

1.3 To determine the clinical relevance of genetic subtyping tumors as a predictor of response to this chemotherapy and long term survival

DETAILED DESCRIPTION:
Capecitabine is a drug that damages the DNA (deoxyribonucleic acid) of tumor cells and blocks the function of DNA and RNA (ribonucleic acid) of tumor cells. These actions help to kill the tumor cells.

Celecoxib is a drug that may help to prevent the development of some types of cancer by blocking a type of enzyme (COX-2) that is found in tumor cells.

Temozolomide and CCNU are the current standard treatment for malignant brain tumors. Both drugs work by damaging the DNA (deoxyribonucleic acid) of tumor cells to kill these tumor cells.

6-Thioguanine is a drug that helps to increase the effects of Temozolomide and CCNU on tumor cells.

Depending on the previous treatment you have received, you will be treated according to Arms 1, 2, or 3.

If you have not received temozolomide before, you will be treated on Arm 1. If you have received temozolomide before but only during radiation therapy and not as chemotherapy afterwards and the treatment was over 6 months ago, you will be treated with temozolomide according to Arm 1.

If you have not received lomustine or carmustine, you will be treated on Arm 2. If you have received Gliadel wafers at surgery greater than 6 months ago and have not been treated with lomustine or carmustine, you will be treated with CCNU according to Arm 2.

Arm 3 will include glioblastoma multiforme patients who may be treated with either temozolomide or lomustine according to the above guidelines and regimens described in Arms 1 and 2.

Arm 1:

Treatment will begin with 6-thioguanine taken by mouth 4 times a day (every 6 hours) for 3 days in a row (Days 1-3). This will be followed by temozolomide taken by mouth at bedtime for 5 days in a row (Days 4-8). After a rest period of 6 days, capecitabine and celecoxib will be taken by mouth twice a day (12 hours apart) for 14 days (Days 14-27). Each cycle of treatment on arm 1 will be 28 days.

Arm 2:

Treatment will begin with 6-thioguanine taken by mouth 4 times a day (every 6 hours) for 3 days in a row (Days 1-3). This will be followed by lomustine taken by mouth at bedtime for 1 day (Day 4). After a rest period of 1 week, capecitabine and celecoxib will be taken by mouth twice a day (12 hours apart) for 14 days (Days 11-24). Each cycle of treatment on arm 2 will take 42 days.

Blood tests (less than 2 teaspoons) will be repeated every 2 weeks and before each new cycle of treatment (a total of about 2 tablespoons). The neurological exam, anticonvulsant level blood tests and the stool test for blood, will be repeated before every cycle on Arms 2 and 3 (CCNU) and before every 2 cycles on Arms 1 and 3 (temozolomide). Kidney function will be evaluated from the blood tests before every other course. Patients taking anticoagulants (coumadin, warfarin) will have procedures to test the clotting ability of the blood before each cycle or more frequently if the doctor feels it is necessary.

Arm 3:

Glioblastoma Multiforme patients will be treated on Arm 3 which will include the drug regimen from either Arm 1 or Arm 2.

Treatment on all arms will continue for 1 year as long as the tumor does not grow and any side effects are tolerable. Treatment may continue beyond one year if your doctor feels it is needed. During the study, you may not receive any other investigational drug or have any other treatment for the cancer, including surgery.

This is an investigational study. All drugs used in this study are FDA approved and are commercially available. A total of 140 patients will take part in this study. All patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital.
2. Patients with histologically proven supratentorial anaplastic oligodendrogliomas, anaplastic mixed oligoastrocytomas anaplastic astrocytomas or glioblastoma multiforme.
3. Patients must have unequivocal evidence for tumor recurrence or progression by MRI scan performed within 14 days prior to enrollment or documented recurrence by tumor resection. Patients must have received radiation therapy previously.
4. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all the following conditions are met: a) Patients have recovered from the effects of surgery; b) Extent of residual disease (if present) has been documented by MRI performed no later than 72 hours after surgery or, if not possible, at least 4 weeks post-operative. Radiographic evidence of residual disease is not mandated for enrollment.
5. The baseline on-study MRI is performed within 14 days of enrollment and on a steroid dosage that has been stable. If the steroid dose is increased between the date of imaging and the initiation of chemotherapy, a new baseline MRI is required on stable steroids for 7 days.
6. Patients must be equal to or greater than 12 years old.
7. Patients must have a Karnofsky performance status of equal to or greater than 60 (Karnofsky Performance Scale; Appendix D).
8. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
9. Patients must have adequate bone marrow function (ANC equal or greater than 1,500/mm3 and platelet count of equal or greater than 100,000/mm3), adequate liver function (SGPT and alkaline phosphatase <2 times normal, bilirubin <1.5 mg%), and adequate renal function (BUN and creatinine <1.5 times institutional normal) prior to starting therapy.

Exclusion Criteria:

1. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years (1 year for localized prostate carcinoma treated by prostatectomy or irradiation) are ineligible.
2. Patients of childbearing potential must not be pregnant or become pregnant.
3. Patients must not have: a) active infection; b) disease that will obscure toxicity or dangerously alter drug metabolism; c) serious intercurrent medical illness; d) acute or chronic pulmonary disease, pulmonary embolus, hypertension, diabetes, metabolic syndrome, stroke, heart disease,myocardial infarction, angina, coronary angioplasty, congestive heart failure, or coronary bypass surgery; e) allergies to sulfa drugs; f) severe psychiatric illness; g) uncontrolled hypertension (i.e. ->135/>85 mm Hg) on three repeated measurements during the 6 weeks prior to enrollment on the study
4. Patients must not have (continued): h) family history of premature coronary disease (i.e. - onset < 55 years of age); i) uncontrolled hypercholesteremia [low-density lipoprotein cholesterol (LDL-C >130]. Hypercholesteremia must be controlled for at least 3 months prior to enrollment on study; j) history of systemic lupus erythematous, family history of protein S or C deficiencies, prior heparin-induced thrombocytopenia, Factor V Leiden deficiencies or high homocysteine levels; k) any indications for ASA deficiency
5. Patients must not have had prior treatment with Capecitabine, 5-FU or a combination of Temozolomide with CCNU (Lomustine) or BCNU (Carmustine). Patients who received only Temozolomide during radiation therapy and did not receive adjuvant chemotherapy with Temozolomide and/or those who received Gliadel (BCNU) wafers at surgery without adjuvant chemotherapy with BCNU or CCNU are eligible if 6 months has passed since the treatment(s).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Conrad, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: U.T. M.D. Anderson's website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 23, 2003 to June 15, 2009. All patients recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Of the 75 enrolled participants, one was excluded prior to assignment to groups. The Anaplastic Tumors Arms (Arm 1 and Arm 2) were combined for recruitment demographics and data collection.
Groups:
- Anaplastic Tumors: 6-TG 80 mg/m^2 orally (PO) every 6 hours Day 1-3; Temozolomide 150 mg/m^2 PO daily Days 4-8 OR Lomustine 100 mg/m^2 PO on Day 4; Capecitabine 825 mg/m^2 every 12 hours; and Celebrex 400 mg PO every 12 hours for 13 days for 28 day course.
- Glioblastoma Multiforme: 6-TG 80 mg/m^2 PO every 6 Hours Day 1-3; Capecitabine 825 mg/m^2 PO every 12 hours Days 14-27 and Celebrex 400 mg PO every 12 hours Day 11-24; Temozolomide 150 mg/m^2 PO daily Days 4-8 OR CCNU (Lomustine) 100 mg/m2 orally Day 4 of each 42-day cycle.
  Participants receive Temozolomide if not had previous treatment and if had prior CCNU. Those previously treated with Temozolomide but not CCNU receive CCNU, and those that had Gliadel and Temozolomide with XRT receive Temozolomide.
Period: Overall Study
Arm/Group | Anaplastic Tumors | Glioblastoma Multiforme
Started | 31 | 43
Completed | 31 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaplastic Tumors | Glioblastoma Multiforme | Total
Number analyzed (Participants) | 31 | 43 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 34 | 63
  >=65 years | 2 | 9 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 17 | 28 | 45
Region of Enrollment [Number; unit: participants]
  United States | 31 | 43 | 74

OUTCOME MEASURES:

1. Primary Outcome: 12 Month-progression-free Survival for Participants With Anaplastic Tumors
Description: Progression-free Survival (PFS) at 12 months measured as percentage of participants that are alive and progression-free at 12 months (anaplastic tumors). A combination of neurological examination and MRI brain scan used to define overall response or progression.
Time Frame: 12 months
Population: Results from TMZ and CCNU treatment arms (Anaplastic Tumor-Glioma Arms 1 & 2) were combined in the final analysis because there was no statistically significant difference between them.
Measure: Number; unit: percentage of participants
Groups:
- Participants With Recurrent Anaplastic Glioma: 6-TG 80 mg/m^2 orally (PO) every 6 hours Day 1-3; Capecitabine 825 mg/m^2 and Celebrex 400 mg PO every 12 hours; Arm 1 Temozolomide (TMZ) 150 mg/m^2 PO daily Days 4-8 OR Arm 2 Lomustine 100 mg/m^2 PO on Day 4; Arm 2 Participants if previously received Temozolomide but not Lomustine (CCNU) receive Lomustine; or if had Gliadel wafers and Temozolomide with radiotherapy (XRT) receive Temozolomide.
Arm/Group | Participants With Recurrent Anaplastic Glioma
Number analyzed (Participants) | 31
percentage of participants | 44 (5)

2. Primary Outcome: 6 Month Progression-free Survival for Participants With Glioblastoma
Description: Progression-free Survival (PFS) at 6 months measured as percentage of participants that are alive and progression-free at 6 months (glioblastoma multiforme). A combination of neurological examination and MRI brain scan used to define overall response or progression.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- Participants With Glioblastoma Multiforme: 6-TG 80 mg/m^2 PO every 6 Hours Day 1-3; Capecitabine 825 mg/m^2 PO every 12 hours Days 14-27 and Celebrex 400 mg PO every 12 hours Day 11-24; Temozolomide 150 mg/m^2 PO daily Days 4-8 OR CCNU (Lomustine) 100 mg/m2 orally Day 4 of each 42-day cycle.
  Participants receive Temozolomide if not had previous treatment and if had prior CCNU. Those previously treated with Temozolomide but not CCNU receive CCNU, and those that had Gliadel and Temozolomide with XRT receive Temozolomide.
Arm/Group | Participants With Glioblastoma Multiforme
Number analyzed (Participants) | 43
percentage of participants | 14

ADVERSE EVENTS:
Time Frame: 6 years and 3 months
Arm/Group | Anaplastic Tumors | Glioblastoma Multiforme
Serious Adverse Events (participants affected / at risk) | 8/31 | 16/43
Other Adverse Events (participants affected / at risk) | 31/31 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaplastic Tumors (N=31) | Glioblastoma Multiforme (N=43)
Thrombosis/Embolism (Vascular disorders) | 1 (1) | 5 (5)
Increased intracranial pressure (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Mental Status (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Hemorrhage (General disorders) | 1 (1) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0)
Pain-Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaplastic Tumors (N=31) | Glioblastoma Multiforme (N=43)
ALKALINE PHOSPHATASE (Metabolism and nutrition disorders) | 5 (6) | 7 (9)
ALLERGIC RHINITIS (Immune system disorders) | 4 (4) | 6 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (8)
ALT SGPT (Metabolism and nutrition disorders) | 10 (13) | 14 (18)
ANEMIA (Blood and lymphatic system disorders) | 6 (16) | 3 (4)
ANOREXIA (Gastrointestinal disorders) | 3 (4) | 5 (5)
AST SGOT (Metabolism and nutrition disorders) | 8 (9) | 10 (13)
BICARBONATE SERUM-LOW (Metabolism and nutrition disorders) | 3 (5) | 4 (12)
BILIRUBIN (Metabolism and nutrition disorders) | 2 (8) | 4 (10)
BLURRED VISION (Eye disorders) | 7 (7) | 9 (13)
BRUISING (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
COGNITIVE DISTURBANCE (Nervous system disorders) | 5 (6) | 5 (5)
CONFUSION (Nervous system disorders) | 5 (6) | 8 (9)
CONSTIPATION (Gastrointestinal disorders) | 15 (32) | 15 (18)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (9)
CREATININE (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 8 (14) | 14 (18)
FATIGUE (General disorders) | 24 (37) | 30 (48)
GAIT/WALKING (Musculoskeletal and connective tissue disorders) | 12 (19) | 13 (18)
HEMOGLOBIN (Blood and lymphatic system disorders) | 24 (60) | 33 (88)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 14 (33) | 43 (47)
HYPERTENSION (Cardiac disorders) | 4 (5) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 7 (11) | 13 (21)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (4) | 10 (18)
HYPONATREMIA (Metabolism and nutrition disorders) | 3 (9) | 9 (10)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 6 (10) | 8 (20)
INSOMNIA (Psychiatric disorders) | 9 (9) | 12 (13)
LEUKOCYTES (Blood and lymphatic system disorders) | 21 (113) | 33 (124)
LEUKOPENIA (Blood and lymphatic system disorders) | 4 (16) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 21 (160) | 33 (147)
MEMORY IMPAIRMENT (Nervous system disorders) | 11 (14) | 18 (20)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 10 (20) | 26 (45)
NAUSEA (Gastrointestinal disorders) | 16 (28) | 16 (26)
NEUTROPHILS (ANC/AGC) (Blood and lymphatic system disorders) | 15 (70) | 28 (72)
PLATELETS (Blood and lymphatic system disorders) | 23 (108) | 31 (96)
PYRAMIDAL TRACT DYSFUNCTION (Nervous system disorders) | 9 (11) | 7 (7)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (7)
SEIZURE (Nervous system disorders) | 10 (14) | 17 (29)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 4 (5) | 3 (4)
VOMITING (Gastrointestinal disorders) | 11 (14) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No